CLINICAL TRIAL: NCT05065840
Title: Implementing an Evidence-Based, Multilevel Intervention to Promote HPV Vaccination Among HIV Positive Adults
Brief Title: Advancing HPV Vaccination Among HIV Positive Adults: The CHAMPS Study
Acronym: CHAMPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jessica Wells, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002469; R01NR020154-01 (NIH)
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Human Papilloma Virus; Human Papilloma Virus Vaccine
Keywords: Human Immunodeficiency Virus; Vaccination
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The study will be implemented at the clinic, Provider, and Patient levels. Every level will receive a different intervention or none in the case of the control. Clinic and Provider level will receive training on recommending and administering the vaccine at the clinic. Patient level will accept or decline the recommendation for the HPV vaccine. The Control arm will be collected from EMR and the GRITS database from patients not receiving the vaccine before the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 Pillars Program (Experimental): Patients at study clinics who consent to have their HPV vaccination history verified with the Georgia Registry of Immunization Transactions and Services (GRITS).
  Interventions: Behavioral: CDC 4 Pillars Program
- Adjacent time-period Control Group (No Intervention): The background HPV update rate among PLWH will be obtained by using the electronic medical record (EMR) and GRITS to identify HPV vaccination uptake 18 months prior to the intervention. These data are collected retrospectively and no study participants are prospectively assigned to this study arm.

INTERVENTIONS:
Behavioral: CDC 4 Pillars Program — The CDC's 4 Pillars Transformation Program (4 Pillars Program) is a robust and empirically supported strategic approach that promotes the uptake of adult vaccinations and addresses facilitators and barriers at the patient, provider, and clinic level. This multi-level, evidence-based intervention has been successfully utilized to increase HPV vaccination in the general population and is primed to be tested in the high-risk HIV population, particularly PLWH in the rural South. This proposal seeks to expand the success of the 4 Pillars Program and tailor, refine, and implement in the HIV positive population who are at extraordinarily high risk for HPV-related cancers and can obtain the most benefit from the vaccine.
  Arms: 4 Pillars Program

SUMMARY:
People living with HIV (PLWH) are 28 times more likely to be diagnosed with Human Papillomavirus (HPV) - associated anal cancer than the general population. The HPV vaccine is an effective and safe approach to prevent and reduce the risk of HPV-related disease among PLWH. HPV vaccine programs tailored and implemented in the HIV population are lagging for this high-risk group. The CDC's 4 Pillars Transformation Program is a multi-level, evidence-based intervention that has been successfully used to increase HPV vaccination in the general population and is ready to be tested in the high-risk HIV population, particularly PLWH in the rural South. This program offers providers and clinic staff evidence-based strategies to increase HPV vaccination uptake via training and educational resources. This study proposes to tailor and refine the 4 Pillars Program and conduct this project in three HIV clinics in Georgia.

DETAILED DESCRIPTION:
People living with HIV (PLWH) are 28 times more likely to be diagnosed with HPV- associated anal cancer than the general population. The HPV vaccine is an effective and safe approach to prevent and reduce the risk of HPV-related disease among PLWH. However, in previous pilot studies, significant gaps were found in knowledge and awareness of the HPV vaccine, as well as low receipt of the HPV vaccine (13.5%) in our population of rural PLWH.

HPV vaccine programs tailored and implemented in the HIV population are lagging for this high-risk group. The Center for Disease Control's (CDC) 4 Pillars Transformation Program is a multi-level, evidence-based intervention successfully used to increase HPV vaccination in the general population and is ready to be tested in the high-risk HIV population, particularly PLWH in the rural South.

The 4 Pillars Program offers providers and clinic staff evidence-based strategies to increase HPV vaccination uptake via training and educational resources. Providers and clinic staff interested in participating will "enroll" online and complete an electronic informed consent before participating in the focus groups and completing the evaluation surveys. Providers and clinic staff will be offered an opportunity to participate in in-service training (CE units will be available) that will provide education and resources on the 4 Pillars program and will learn more about HPV, HPV vaccination, and HPV-associated cancers. Providers and clinic staff will be asked to recommend and administer the HPV vaccine during each routine clinic visit. Consenting providers and clinic staff will be asked to complete pre-intervention evaluations, an intervention evaluation every 3 months, a post-evaluation, and post-intervention assessments.

For patient enrollment, the research coordinator, with assistance from a clinic-designated Immunization Champion (IC), will review the clinic's appointment schedule to call patients in the target age range (18- 45 years of age) one week in advance of their appointments to inform them of the study and to determine eligibility. If eligible and interested in the proposed study, the individual will be given an overview of the research study, including its purpose, what participation entails, potential risks and benefits of participation, and measures that will be used to ensure confidentiality. Participants will be assured that participation is completely voluntary, and they may withdraw from the study at any time without consequences. If the individual volunteers to participate in the study, an electronic informed consent will be obtained by the research assistant(s) via REDCap. Participants will be asked to consent to have their HPV vaccination status confirmed via electronic medical records and GRITS. Participants will then watch a short video on HPV and HPV vaccines that can be viewed on their phones (or the clinic's iPad) while waiting to be seen. Potential participants will be asked to "follow" the study's private Facebook page, which will offer additional educational information tailored towards individuals with HIV on HPV-related disease and general health promotion and risk reduction tips. A post-intervention evaluation will be provided after the third immunization is given or due (if missed).

ELIGIBILITY:
Inclusion Criteria

* HIV positive
* 18-45 years of age
* Can read and speak English
* Capable of providing informed consent
* Has not previously received three series HPV vaccine
* No contraindications to receiving HPV vaccine (i.e. history of anaphylactic allergy to later, an immediate hypersensitivity to yeast, current moderate or severe acute illness, and/or are currently pregnant).

Exclusion Criteria:

* Has contraindications to receiving the HPV vaccine i.e., history of an anaphylactic allergy to latex, an immediate hypersensitivity to yeast, current moderate or severe acute illness, and/or are currently pregnant)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 365 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients initiating the HPV vaccine | 24 months post baseline
  Initiation of the HPV vaccine is defined as receiving the first or second immunization from the series. This variable will be measured by electronic medical records and GRITS at 24 months post baseline.

SECONDARY OUTCOMES:
Number of participants completing the HPV vaccine | 24 months post baseline
  Completion is defined as receiving all 3 immunizations from the series, regardless of time. This variable will be measured by electronic medical records and GRITS 24 months post baseline.
Change in uptake rate of vaccination | Baseline and 24 months post baseline
  The team will calculate the percent change in initiation of the vaccine and percent change in completion of the vaccine from the control phase and 24 months post intervention, after adjusting for demographics differences in population.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Wells, PhD, RN, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Albany Rural Model Clinic, Albany, Georgia
  - AID Atlanta, Atlanta, Georgia
  - Faebris, Atlanta, Georgia
  - AHF Lithonia, Lithonia, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual data that underlie the results of the study's specific aims. All reported data, including text, tables, figures, and appendices, will be de-identified.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee, for individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata

REFERENCES:
- [Derived] Wells J, Klosky JL, Liu Y, Gillespie TW. An overview of implementing an evidence based program to increase HPV vaccination in HIV community clinics. BMC Public Health. 2022 Sep 7;22(1):1696. doi: 10.1186/s12889-022-14100-0. PMID 36071389